CLINICAL TRIAL: NCT06754956
Title: Imaging Study of Intracranial and Extracranial Arterial Atherosclerotic Plaques Using 3.0T and 5.0T MRI: A Prospective Self-Controlled Study
Brief Title: Imaging of Intracranial and Extracranial Arterial Atherosclerotic Plaques Using Different Field Strength MRIs
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Jiao Tong University Affiliated Sixth People's Hospital (Other)
Responsible Party: Principal Investigator, Yueqi Zhu, MD, Shanghai Jiao Tong University Affiliated Sixth People's Hospital
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: Imaging-SISTER study
Record Dates: First submitted 2024-12-24; First posted 2025-01-01 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: High Resolution Vessel Wall Imaging; Intracranial Atherosclerotic Stenosis, ICAS; Arteriosclerosis
MeSH Terms: conditions — Splenic Hypoplasia; Arteriosclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patients underwent both 3.0T and 5.0T HR-VWI MRI (Experimental)
  Interventions: Device: The patient will receive two intravenous injections of the same gadoterate meglumine contrast agent.

INTERVENTIONS:
Device: The patient will receive two intravenous injections of the same gadoterate meglumine contrast agent. — Each patient will undergo two different field strength HR-VWIs with enhancement, and on each occasion the patient will be injected with contrast DOTAREM (gadoterate meglumine) .

SUMMARY:
Atherosclerotic stenosis of the carotid and intracranial arteries is one of the leading causes of ischemic cerebrovascular events worldwide. Among these, intracranial atherosclerotic stenosis has an incidence rate of up to 46.6% in patients with ischemic stroke or transient ischemic attack (TIA) in China. The continuous advancement of high-resolution vascular wall imaging (HR-VWI) technology has enabled multi-dimensional imaging of the arterial walls of both intracranial and extracranial vessels. By suppressing intravascular flow, this technique allows clear visualization of the vascular wall morphology and signal characteristics, as well as the identification of plaque composition and assessment of vulnerable plaque features. However, due to the smaller size of intracranial atherosclerotic plaques, the image quality and effectiveness of current 3.0T high-resolution magnetic resonance imaging (MRI) are influenced by hardware and software limitations, as well as imaging parameters, making it difficult to accurately perform qualitative and quantitative analysis of intracranial and extracranial plaques. The advent of ultra-high field 5.0T MRI overcomes the limitations of 3.0T MRI in imaging, significantly improving the signal-to-noise ratio and allowing for clearer visualization of the signal characteristics of the arteria.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years;
* Moderate to severe intracranial or extracranial arterial stenosis (stenosis degree: 50% to 99%, confirmed by CTA, MRA, or DSA);
* Written informed consent signed by the patient or their legal representative.

Exclusion Criteria:

* Non-atherosclerotic intracranial arterial stenosis, such as dissection or moyamoya disease;
* Contraindications to MRI, such as claustrophobia or presence of a cardiac pacemaker;
* Allergy to gadolinium-based contrast agents;
* Poor MRI image quality preventing analysis;
* Abnormal liver or kidney function;
* History of any prior endovascular treatment;
* Presence of implants posing potential safety risks in 5.0T MRI, such as non-removable metallic dental prostheses, stents, or other metallic implants.

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-01-10 (Actual); Primary Completion 2027-09-23 (Estimated); Study Completion 2027-12-23 (Estimated)

PRIMARY OUTCOMES:
Comparison of the Accuracy of Clinical Event-Based Definition of Plaque Vulnerability Assessed by 5.0T and 3.0T HR-VWI. | immediately after HR-VWI injection

SECONDARY OUTCOMES:
Comparison of image quality of 5.0T and 3.0T HR-VWI. | immediately after HR-VWI injection
Comparison of clinicians' visual scale for 5.0T and 3.0T HR-VWI. | immediately after HR-VWI injection
  The clinicians' visual scale is a four-point scale. 1 for inadequate, 2 for adequate, 3 for good, 4 for excellent. In detail, excellent rated images meant clear vessel wall delineation for entire boundary. Good images showed good vessel wall delineation with only small part of obscure/invisible boundary. Adequate rated images stood for reasonable image quality on vessel wall visualization involving some part but less than a quadrant of obscure/invisible boundary. Inadequate images were those in which most of the vessel wall boundaries could not be seen.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Sixth People's Hospital, Shanghai,200023, Shanghai, China

IPD SHARING:
Plan to Share IPD: No